CLINICAL TRIAL: NCT02615626
Title: Gingival Crevicular Fluid and Serum Levels of Visfatin in Periodontal Diseases Before and After Non-surgical Periodontal Treatment
Brief Title: Visfatin Levels Before and After Periodontal Treatment
Acronym: VL
Status: Completed | Type: Observational
Sponsor: Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, ÇİĞDEM COŞKUN TÜRER, Dr, Bulent Ecevit University
Other Study IDs: VLandPT
Record Dates: First submitted 2015-11-23; First posted 2015-11-26 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-11

CONDITIONS: Periodontal Diseases
Keywords: Visfatin; GCF; serum; Non-surgical Periodontal Treatment.
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Gingival crevicular fluid and Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group 1: Periodontal healthy
  Interventions: Procedure: Non-surgical Periodontal Treatment.
- Group 2: Gingivitis, Non-surgical Periodontal Treatment
  Interventions: Procedure: Non-surgical Periodontal Treatment.
- Group 3: Chronic Periodontitis, Non-surgical Periodontal Treatment
  Interventions: Procedure: Non-surgical Periodontal Treatment.

INTERVENTIONS:
Procedure: Non-surgical Periodontal Treatment. — Non-surgical periodontal therapy is an anti-infective therapy which includes both mechanical and chemotherapeutic approaches to minimize or eliminate microbial biofilm, the primary etiology of gingivitis and periodontitis

SUMMARY:
The purpose of this study was to evaluate visfatin levels in different stages of periodontal diseases and health, moreover the effect of non-surgical periodontal therapy on visfatin levels in Gingival Crevicular Fluid (GCF) and Serum.

DETAILED DESCRIPTION:
Total of 45 patients were divided into three groups based on their clinical and radiographical examination. Group 1 chronic periodontitis (n: 15), group 2 plaque induced gingivitis (n: 15) and group 3 Periodontal health (n: 15). GCF and serum samples were collected before treatment and 1, 3, 6 months after treatment and were assayed using enzyme linked immunosorbent assay kit.

ELIGIBILITY:
Group 1 Inclusion Criteria:

* GI>1, PPD≥5mm, CAL≥5mm with alveolar bone loss radiographically.
* Systematically healthy patients

Group 2 Inclusion Criteria:

* No alveolar bone and attachment loss
* Inflammation signs such as redness, edema and increased BOP levels,
* GI≥2, PPD≤3mm, CAL≤3mm.
* Systematically healthy patients

Group 3 Inclusion Criteria:

* No bone and attachment loss,
* GI=0, PPD≤3mm, CAL≤3mm
* Systematically healthy patients

Exclusion Criteria for all groups:

* Aggressive Periodontitis,
* Oral pathologies,
* Patients with any other systemic diseases,
* Pregnant women and those in the lactation period,
* Patients with smoking habit and taking medication
* Patients received periodontal therapy in last 6 months

Ages: 25 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Total of 45 patients
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2012-05; Primary Completion 2013-10 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Visfatin levels: Change after periodontal treatment both in serum and GCF | baseline, 1, 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: ÇİĞDEM COŞKUN TÜRER, Ph.D, Principal Investigator — BULENT ECEVIT UNIVERSITY FACULTY OF DENTISTRY DEPARTMENT OF PERIODONTOLOGY